CLINICAL TRIAL: NCT03271996
Title: Two Surgical Techniques for the Treatment of Pilinidal Sinus: A Randomized Controlled Trial
Brief Title: Fistulectomy vs. Modified Karydakis Procedure for Pilonidal Sinus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Dimitri Christoforidis (Other)
Responsible Party: Sponsor-Investigator, Dimitri Christoforidis, Vice-Chief in Surgery, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-016
Record Dates: First submitted 2017-08-17; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Pilonidal Sinus
Keywords: Pilonidal sinus; Bascom; Cleft lift; Fistulectomy; Karydakis
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary closure (Experimental): Excision of sinus and paramedian closure according to modified Karydakis technique
  Interventions: Procedure: Primary closure
- Fistulectomy (Experimental): Removal / fistulectomy by scalpels or trephines of primary and drainage orifices and healing of the wound by second intention
  Interventions: Procedure: Fistulectomy

INTERVENTIONS:
Procedure: Primary closure — Asymmetric skin incision and total excision of the lesion with monopolar scalpel. Accurate hemostasis, creation of a cutaneous-subcutaneous flap, primary closure with non-absorbable sutures, optional aspiration drainage.
  Arms: Primary closure
Procedure: Fistulectomy — Evaluation of the cavity using a 0.5-1 mm metal probe which will be inserted into the skin orifice. Excision of the skin around the orifice and debridement/excision of the cavity by monopolar scalpel or Trephines
  Arms: Fistulectomy

SUMMARY:
This study wants to improve patient care affected by pilonidal sinus during and after surgery. Pilonidal sinus excision is a frequent procedure, despite this, there is still not an appropriate surgical technique because of a lack of quality comparative studies.

DETAILED DESCRIPTION:
This is a randomized controlled trial. The study will compare the healing of the surgical wound and the recurrence rate after excision and primary para-median closure versus narrow orifice excision (fistulectomy)

Group A: excision and paramedian closure according to modified Karydakis technique

Group B: removal / fistulectomy by scalpels or trephines of primary and drainage orifices, healing of the wound by secondary intention

ELIGIBILITY:
Inclusion Criteria:

* Pilonidal cyst requiring surgery
* Signed Informed Consent Form

Exclusion Criteria:

* Abnormal lesions
* Injuries requiring a closing with rotation flap

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Complete healing | 3 weeks
  percentage of complete healing

SECONDARY OUTCOMES:
Time to recovery | 12 months
  Time to completely recovery
percentage of relapse | 12 months
  percentage of relapse after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Regionale di Lugano, Lugnao, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Popeskou SG, Pravini B, Panteleimonitis S, Vajana AFDT, Vanoni A, Schmalzbauer M, Posabella A, Christoforidis D. Conservative Sinusectomy vs. excision and primary off-midline closure for pilonidal disease: a randomized controlled trial. Int J Colorectal Dis. 2020 Jul;35(7):1193-1199. doi: 10.1007/s00384-020-03551-9. Epub 2020 Mar 6. PMID 32144531